CLINICAL TRIAL: NCT02842125
Title: Phase 1/2 Evaluation of Adenoviral p53 (Ad-p53) in Combination With Capecitabine (Xeloda) or Anti-PD-1 in Patients With Unresectable Liver Metastases of Colorectal Carcinoma(CRC) and Other Solid Tumors, Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC) and Primary Hepatic Cancers With Known Disease Progression on Standard Therapy
Brief Title: Safety and Efficacy of Intra-Arterial and Intra-Tumoral Ad-p53 With Capecitabine (Xeloda) or Anti-PD-1 in Liver Metastases of Solid Tumors and Recurrent Head and Neck Squamous Cell Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Arm C rolled into parallel study; Arms A and B halted for greater efficacy in Arm C
Sponsor: MultiVir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MultiVir Ad-p53-001
Record Dates: First submitted 2016-07-01; First posted 2016-07-22 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Solid Tumor Cancer; Recurrent Head and Neck Cancer
Keywords: Head and Neck Squamous Cell Cancer; solid tumors; nivolumab; Ad-P53; metastatic; capecitabine; pembrolizumab
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis | interventions — advexin; Capecitabine; pembrolizumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: 3 Arms, no cross-over
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ad-p53 with Xeloda 33.3% of patients (Experimental): Up to 12 patients, in 3+3 cohorts, all patients treated with Intra-arterial Ad-P53 once weekly, dosing dependent on DLT and MTD findings, and daily metronomic Xeloda (capecetabine), at a dose of 625 mg/m2 BID continuously.
  Interventions: Drug: Ad-P53; Drug: Xeloda
- Ad-p53 with Keytruda 33.3% of patients (Experimental): Up to 12 patients, in 3+3 cohorts, all patients treated with Intra-arterial Ad-P53 once weekly, dosing dependent on DLT and MTD findings, and infusions of pembrolizumab every 3 weeks.
  Interventions: Drug: Ad-P53; Drug: Keytruda
- Ad-p53 with Opdivo 33.3% of patients (Experimental): Up to 12 patients treated with intra-tumoral Ad-P53 3 times week 1 of each cycle, dose determined by tumor size, in combination with IV nivolumab (Opdivo) 480 mg, every 4 weeks.
  Interventions: Drug: Ad-P53; Drug: Opdivo

INTERVENTIONS:
Drug: Ad-P53 — Adenoviral Investigational Product Ad-P53 to treat metastases using an intra-arterial catheter, with oral metronomic capecitabine
Drug: Xeloda — Oral metronomic chemotherapeutic agent
  Other Names: capecitabine
  Arms: Ad-p53 with Xeloda 33.3% of patients
Drug: Keytruda — Antineoplastic, Monoclonal Antibody; PD-1/PD-L1 Inhibitors
  Other Names: Pembrolizumab
  Arms: Ad-p53 with Keytruda 33.3% of patients
Drug: Opdivo — Antineoplastic, Monoclonal Antibody; PD-1/PD-L1 Inhibitors
  Other Names: Nivolumab
  Arms: Ad-p53 with Opdivo 33.3% of patients

SUMMARY:
This is a Phase 1/2 study of the combination of Ad-p53 administered intra-arterially in combination with oral metronomic capecitabine or pembrolizumab in patients with unresectable, refractory liver metastases of colorectal carcinoma (CRC) and other solid tumors, including primary hepatocellular carcinoma (HCC). A third arm will study the intra-tumoral injection of Ad-p53 combined with nivolumab infusions in recurrent head and neck squamous cell cancer (HNSCC). This safety study has a standard 3+3 design for arms A and B; .HNSCC will be placed in a single dosing cohort. The Maximum Tolerated Dose (MTD) will be determined as well for intra-arterial infusions, and the entire study will determine the general efficacy using RECIST 1.1 and Immune-Related Response Criteria. Safety will be followed using the CTCAE listings for adverse events.

DETAILED DESCRIPTION:
This is a Phase 1/2 study split into 3 arms. Arm A will follow the combination of Ad-p53 administered intra-arterially in combination with oral metronomic capecitabine while Arm B follows the intra-arterial administration of Ad-p53 combined with pembrolizumab, both in patients with unresectable, refractory liver metastases of colorectal carcinoma (CRC) and other solid tumors, including primary hepatocellular carcinoma (HCC). Arm C will follow the combination of intra-tumoral injections of Ad-p53 and nivolumab infusions. Arms A and B have a standard 3+3 design, with dosing following the initial cohort determined by MTD and DLT criteria as well as safety and tolerance. Arm C will be a single dosing cohort followed for safety and efficacy. All patients will be followed for adverse events and preliminary efficacy. In Arms A and B, the Maximum Tolerated dose (MTD) will be determined. All patients will be followed for general safety and preliminary efficacy using RECIST 1.1 and Immune-Related Response Criteria. CEA levels will also be followed for patients with metastatic colo-rectal cancer. Biomarker testing of archival or fresh tissue is performed during the study. In Arms A and B, patients will undergo a maximum of 2 8-week cycles, with scans every 8 weeks. For Arm B, patients will undergo a maximum of 3 28-day Cycles. All patients will continue on the background therapy for any additional cycles. No additional biopsies are planned following Screening. Enrollment will be up to 24 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male or female, age 18 or above, who agree to use barrier contraception throughout the study. Females of child-bearing potential must be non-pregnant and non-lactating throughout the study.
3. Histologically or cytologically confirmed solid tumors or hepatocellular carcinoma with known disease progression.
4. Each patient entered on the study must have disease that is evaluable for response using RECIST 1.1 criteria with a minimum size of 1 cm by CT/MRI or physical examination
5. Carcinoma patients in Arm A or Arm B must have received at least 1 prior regimen of standard of care systemic antitumor therapy for their metastatic disease and experienced tumor progression within 3 months after the last prior administration of the therapy or experienced unacceptable toxicity to these treatments.
6. Subjects in Arm A and Arm B should have measurable CT evidence of liver metastases or liver lesions that are not treatable by surgical resection or local ablation in consultation with hepatobiliary specialist.
7. The maximum tumor diameters for each Cohort for both Arm A and Arm B should achieve a dose of approximately 1x1011 viral particles (vp)/cm3 of tumor volume. (see Table 1). Please refer to Table for calculating tumor volume.
8. ECOG Performance Status 0 - 1
9. Either no brain metastases or irradiated stable brain metastases
10. Life expectancy at least 3 months
11. No prior autologous or allogeneic organ or tissue transplantation
12. PT/international normalized ratio (INR) ≤ULN; aPTT ≤ULN.
13. ANC ≥1500 cells/mm3
14. Platelet count ≥100,000 cells/mm3
15. Hemoglobin ≥9.0 g/dL
16. Creatinine <2.0 mg/dL or creatinine clearance ≥50 mL/min
17. Total bilirubin <1.5 x ULN
18. AST and ALT <3.0 x ULN
19. Alkaline phosphatase ≤5 x ULN
20. Negative pregnancy test in women of childbearing potential
21. Fertile patients must use effective contraception
22. No non-approved investigational agents or procedures ≤4 weeks of study entry
23. Patients with PRIMARY HEPATIC CANCER must have an undetectable viral load for Hepatitis B and C.
24. Patients with Primary Hepatic Cancer have not recently been treated with antivirals.
25. Troponin blood level within normal limits.
26. Favorable biomarker profile defined by either wild type p53 gene sequence or less than 20% p53 positive tumor cells by immunohistochemistry
27. Echocardiogram with normal ejection fractions
28. Normal lung oxygen saturation by pulse oximeter, as determined by the Principal Investigator based on patient history and status.
29. Arm C patients must have loco-regional recurrent head and neck squamous cell carcinoma (HNSCC), excluding endolaryngeal recurrence, meeting the following criteria:

    * Tumor progression within 6 months of platinum-based chemotherapy
    * All HNSCC lesions should be in the head and neck region and suitable for intra-tumoral injection
    * The total sum of Ad-p53 Injection Doses (mL) based upon the tumor volumes shown in Table 2 should be less than or equal to 25 mL as the MTD of Ad-p53 is 2.5 x1013 vp/treatment day.

Exclusion Criteria

1. Subjects must not be candidates for hepatic surgery or locoregional therapy of liver tumors with curative intent.
2. Liver tumors must not be estimated to invade approximately more than one-third of the liver.
3. Liver tumor-directed therapy, hepatic surgery, antibody-based therapy, or immunotherapy must not have been performed < 28 days, chemotherapy < 21 days, and targeted small molecule therapy or hormonal therapy < 14 days prior to enrollment. No radiation to tumor sites during the last 4 weeks.
4. No macroscopic intra-vascular invasion by tumors of the main portal vein, hepatic vein or vena cava.
5. Chronic liver dysfunction prior to development of liver metastases (Child-Pugh C or greater).
6. Active alcohol dependence
7. Prior radiation performed to areas of measurable disease ≤ four weeks of study entry unless there is documented evidence of disease progression.
8. Use of systemic anti-cancer therapy ≤ 4 weeks, or six weeks if the systemic therapy contains a nitrosourea or mitomycin C.
9. Neuropathy (≥grade 2 CTCAE)
10. History of allergic reactions to any components of the treatments
11. Prior additional malignancy within 2 years except for non-melanoma skin cancer, carcinoma in situ of the breast, oral cavity or cervix.
12. Severe, active comorbidity, including any of the following:

    1. Active clinically serious infection requiring intravenous antibiotics at the time of study entry (CTCAE Grade 2)
    2. Hepatic insufficiency not due to tumor resulting in clinical jaundice or bilirubin >1.5 x ULN and/or coagulation defects
    3. Thrombotic or embolic event within the last 6 months including portal vein thrombosis
    4. Must not require concomitant treatment with anticoagulants
    5. QTcb >470 ms
    6. Bleeding or evidence or history of clinically significant bleeding diathesis or coagulopathy within the last 3 months
    7. Uncontrolled hypertension on anti-hypertensive medication (systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg)
    8. Must not have been diagnosed with autoimmune disease or be immunosuppressed
    9. Patients with non-hepatocellular carcinoma must not have acute or chronic hepatitis B or hepatitis C infection
    10. Known significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or immunosuppressive medication including high-dose corticosteroids.
    11. Severe bleeding, hemoptysis, gastrointestinal hemorrhage, CNS bleeding, clinically significant hemorrhage or vaginal bleeding during the last 6 months
    12. Subjects must not have evidence of pneumonitis or inflammatory lung disease on CT scan and x-ray
13. Chronic treatment for more than 6 months with systemic corticosteroids at doses above 10 mg prednisolone or equivalent before study entry
14. Psychological, familial, sociological or geographical or other condition which in the opinion of the investigator would not permit study follow-up or other compliance with the study protocol.
15. Subjects must not have tumors adjacent to vital structures such as carotid arteries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Safety assessed by CTCAE | Screening to 30-days following Final Treatment (approximately 22 weeks)
  Incidence of treatment-emergent and treatment-related adverse events (all AEs, laboratory AEs, SAEs and Fatal AEs, in accordance with the CTCAE
Incidence of dose-limiting toxicities (DLTs) | Day 1 to 30-days Following Last Treatment (approximately 21 weeks)
  To evaluate the safety, as assessed by the incidence of dose limiting toxicities, of the combination of Ad-P53 and Xeloda or Ad-p53 and Keytruda
Determination of maximum-tolerated dose (MTD) | Day 1 to 30 days following Final Treatment (Approximately 21 Weeks)
  Determination of maximum tolerated dose (MTD) by review of DLTs, of the combination of Ad-p53 and Xeloda or Ad-p53 and Ketruda
Progression-Free Survival (PFS) of patients using RECIST 1.1 | Time Frame: Day 1 to progression through end of study, approximately 18 months
  PFS in patients treated with Ad-p53 and nivolumab determined by review of scans every 8 weeks for disease progression in accordance with RECIST 1.1. Scans are read locally but kept for possible central review. Scans are done every 8 weeks. Sites will review questionable findings on scans with Immune Related Response Criteria (irRC) [Wolchok 2009].

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) of patients using RECIST 1.1 | Day 1 to progression through end of study, approximately 2 years
  PFS determined by review of scans every 8 weeks for disease progression in accordance with RECIST 1.1 in patients treated with Ad-p53 and either Xeloda or Keytruda. Scans are read locally but kept for possible central review. Scans are done every 8 weeks.
Efficacy determined by Immune Related Response Criteria (irRC) [Wolchok 2009] | Day 1 of Treatment through 30-days following last treatment (20 weeks)
  Efficacy will be determined by review of the irRC (Immune-Related Response Criteria. Patients will undergo scanning every 8 weeks for the duration of the study, with evaluation of the scans in accordance with the Immune Related Response Criteria, including confirmation of disease progression with a scan 4 weeks after noted per RECIST criteria.
Efficacy as determined by biomarker testing and immunohistochemistry testing | Day 1 of Treatment to End of Study (approximately 18 months)
  Efficacy endpoints will be correlated with central biomarker testing for PDL-1, PD-2, as well as central biomarker testing for immune cell infiltrates and tumor mutational burden biomarkers in exploratory analyses, through Cancer Genetics, Inc.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Subbiah, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No